CLINICAL TRIAL: NCT03843294
Title: Phase I Study Utilizing Tumor Associated Antigen Specific T Cells (TAA-T) With PD1 Inhibitor Nivolumab for Relapsed/Refractory Lymphoma
Brief Title: Tumor Associated Antigen Specific T Cells (TAA-T) With PD1 Inhibitor for Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Bollard (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Director - Center for Cancer and Immunology Research, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUSTAIN
Record Dates: First submitted 2019-01-16; First posted 2019-02-18 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab with TAA-T cell (Experimental): Patients will receive doses of Nivolumab at a minimum of 8 weeks prior to first TAA-T cell infusion and additional dose(s) of Nivolumab will be given after 4 weeks following second TAA-T cell infusion starting at week 7 from first infusion of TAA-T.If patient meets eligibility criteria for TAA-T cell infusion, the patient will receive two TAA-T cell infusions given 2 weeks apart
  Interventions: Biological: TAA-T cells; Drug: Nivolumab

INTERVENTIONS:
Biological: TAA-T cells — The patient will receive two TAA-T cell infusions given 2 weeks apart. TAA-T cell dose: 2 x 107 cells/m2.per infusion.
Drug: Nivolumab — Nivolumab: For patients <18 years, 3 mg/kg/dose (maximum 240mg/dose) every 2 weeks. For adult patients ≥18 years, a dose of 240mg every 2 weeks or 480mg every 4 weeks

SUMMARY:
This is a Phase I, open-label multi-site trial designed to evaluate the safety of administering rapidly-generated Tumor associated antigen specific T cells (TAA-T) with the Programmed Death1 (PD-1) inhibitor Nivolumab, in relapsed/refractory lymphoma (rel/ref) patients with measurable disease (group A) or as adjunctive therapy following autologous hematopoeitic stem cell transplant(HSCT) for patients at high risk of relapse (group B).

The purpose of this study is to find out if the tumor specific T cells given with Nivolumab are safe and to learn what the side effects are and if the combination can help patients with relapsed lymphomas.

DETAILED DESCRIPTION:
This Phase I, open-label multi-site trial is designed to evaluate the safety of administering rapidly-generated multi-antigen-specific T lymphocytes with the PD1 inhibitor Nivolumab, to relapsed/refractory (rel/ref) lymphoma patients with measurable disease (group A) or as adjunctive therapy following autologous HSCT (group B).

This study will first enroll 6 patients total (in Groups A and B) in the initial safety monitoring or DLT group prior to the expansion phase where additional 12 patients (6 in Group A and 6 in Group B) will be enrolled. TAA-T cells will be generated from patient's lymphocytes obtained from patient's PBMC.

If patient meets eligibility criteria for TAA-T cell infusion, the patient (Group A or Group B) will receive two TAA-T cell infusions given 2 weeks apart, where the expected volume of infusion is 1 to 10 cc.

Both TAA-T cells and Nivolumab will be given at the doses below with allowed de-escalation of both doses as follows:

* TAA-T cell dose: 2 x 107 cells/m2 per infusion
* Nivolumab: For patients <18 years, 3 mg/kg/dose (maximum 240mg/dose) every 2 weeks. For adult patients ≥18 years, a dose of 240mg every 2 weeks or 480mg every 4 weeks

From the first 2 enrolled patients, if at least one patient meets dose limiting toxicity criteria (as described in section 6.4.1) at the above mentioned combination dose level, then the next 2 patients will receive TAA-T cells at 1 x 107 cells/m2 without a change in Nivolumab dose. If toxicity criteria are met by at least one patient from these 2 patients, then the dose of Nivolumab will be reduced to 1mg/kg/dose for patients <18 years or 100mg if receiving 240mg dosing or 200mg if receiving 480mg dosing for adult patients ≥18 years for next 2 patients and TAA-T cells will be given at the same de-escalated dose of 1x 107 cells/m2.

In case the patient experiences toxicity from Nivolumab prior to the first TAA-T cell infusion, they can receive the TAA-T cells after resolution of the Nivolumab toxicities and steroid dosing has been reduced less than 0.5mg/kg/day.

After the safety phase is complete, additional 12 patients total will be enrolled on expansion cohort.

Patients will receive doses Nivolumab at a minimum of 8 weeks prior to first TAA-T cell infusion and additional dose(s) of Nivolumab will be given after 4 weeks following second TAA-T cell infusion starting at week 7 from first infusion of TAA-T.. Delays >3 days for the Nivolumab will not be considered protocol violations if discussed with the PI.

If the TAA-T cells are not ready after the initial doses of Nivolumab prior to the first TAA-T infusion, then the patients can continue Nivolumab infusions for an additional 8 weeks at the PI's discretion. If there is insufficient number of TAA-Ts for the two planned infusions, then additional blood may be drawn and patients can continue on Nivolumab unless they rapidly progress with disease requiring urgent therapy. If there is insufficient number of TAA-Ts to meet study dose, a lower dose of TAA-T may be infused at the discretion of the PI.

Only group A patients are eligible for additional doses ( 3 to 8) if they have stable disease or response, do not have ≥ grade 3 toxicity attributed to TAA-T cells and do not have clinical evidence of rapidly progressing disease requiring urgent therapy.

For Group B patients, blood for generation for TAA-T cells (non-mobilized) will be collected prior to the stem cell collection or any time after Day 30 post auto-HSCT. Treatment with Nivolumab will begin any time after Day 30 post auto-HSCT. Patients are eligible for Group B if they have no evidence of metabolically active disease by PET/CT (Deauville Score of 3 or less) at time of starting treatment with Nivolumab. Patients eligible for Group B with <CMR)/CR (by PET/CT) prior to auto-HSCT will need to be in CR (Deauville Score of 3 or less) prior to the start of Nivolumab or can be moved to Group A if they have metabolically active disease (Deauville Score of 4 or more) by PET/CT.

Patients should not receive other systemic antineoplastic agents including Nivolumab for at least 6 weeks after the first infusion of TAA-specific T-cells (for purposes of evaluation), although such treatment may be added if deemed critical for patient care by the attending physician.

Patients in Group A will not be able to receive additional doses (3-8) of TAA-T cells until the initial 6 weeks evaluation for toxicity and efficacy following the first TAA-T cell infusion.

Patients (Group A and B) will not receive subsequent doses of Nivolumab until the safety evaluation for TAA-T is over (at least 6 weeks from the first infusion).

ELIGIBILITY:
Disease Specific Inclusion Criteria

Group A (patients with measurable disease) Relapsed/Refractory Hodgkin Lymphoma (HL) and Diffuse Large B cell Lymphoma (DLBCL) DLBCL

* Patients who have failed at least 2 lines of prior therapy with a failed attempt at both an autologous stem cell transplant and chimeric antigen receptor T cell therapy.
* Patients who are deemed autologous stem cell transplant ineligible and have failed only one line of prior therapy.
* Systemic therapies to treat prior indolent lymphomas count towards previous DLBCL lines of therapy unless the treatment was anti-CD20 antibody monotherapy.

HL

* Rel/ref HL failing more than or equal to 1 salvage regimens, including prior Brentuximab Vedotin (BV)
* Rel/ref after autologous HSCT

Group B (consolidation after auto-HSCT for patients at high risk for relapse) DLBCL

* Patients with < CMR/CR (by PET/CT) with initial treatment regimen
* Patients with relapse <12 months from diagnosis or <6 months from completion of initial therapy
* Patients with <CMR/CR (by PET/CT) prior to autologous HSCT
* Patients requiring >1 salvage regimen prior to autologous HSCT HL
* Patients with relapse <12 months from diagnosis or <6 months from completion of initial therapy
* Patients with <CMR/CR (by PET/CT) prior to autologous HSCT
* Patients requiring >1 salvage regimen prior to autologous HSCT

Recipient Inclusion Criteria for Initial and Subsequent Procurements (TAA-T Cell Generation):

* Age >12 years
* Karnofsky/Lansky score of more than or equal to 50 (see appendix C).
* ALC > 600
* Patients receiving Granulocyte colony-stimulating factor (G-CSF) are recommended a washout period of a minimum of two weeks before procurement
* Agree to use contraceptive measures during study protocol participation (when age appropriate)
* Patient or parent/guardian capable of providing informed consent

Recipient Exclusion Criteria for Initial and Subsequent Procurements (TAA-T Cell Generation):

* Prior allogeneic BMT
* Prior solid organ transplant
* Patient who has received ATG, Campath or other immunosuppressive T cell monoclonal antibodies within 28 days of screening for enrollment
* Patient with uncontrolled infections
* Patient with active HIV
* Pregnancy or lactating
* Failure to meet institutional guidelines for treatment with Nivolumab

Recipient Inclusion Criteria for Initial and Subsequent TAA-T Cell Infusions:

* Age >12 years
* Patient has received at least 8 weeks of Nivolumab
* Patients with Grade 1 toxicities attributed to Nivolumab will be eligible at the discretion of the PI. Toxicities include but not limited to: laboratory abnormalities in thyroid function tests suggestive of hypothyroidism, thyroiditis or thyroid dysfunction adequately managed with thyroid hormone replacement, or abnormalities in amylase, lipase
* Steroids less than 0.5 mg/kg/day prednisone or equivalent
* Karnofsky/Lansky score of more than or equal to 50
* Pulse oximetry of > 90% on room air
* Bilirubin less than or equal to 2.5 mg/dL, AST/ALT less than or equal to 5x upper limit of normal, serum creatinine < 1.0 or 2x the upper limit of normal (whichever is higher)
* Absolute neutrophil count > 250/µL (may be supported with GCSF)
* Agree to use contraceptive measures during study protocol participation (when age appropriate)
* Patient or parent/guardian capable of providing informed consent

Recipient Exclusion Criteria for Initial and Subsequent TAA-T Cell Infusions:

* Investigational therapies within 28 days prior to screening for enrollment
* Uncontrolled infections
* Patient with ≥ grade 1 or symptomatic non-hematologic toxicities from prior therapies

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Product-Emergent Adverse Events | 6 weeks from the first TAA-T cell administrations
  Number of participants with grades 3-5 infusion-related and grades 4-5 non-hematological adverse events that are not due to the original malignancy, or pre-existing co-morbidities at least 6 weeks of the first dose of TAA-T infusion as defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03, change from baseline up to week 6.

SECONDARY OUTCOMES:
Tumor response to combination immunotherapy | 1 year
  Number of patients with tumor associated antigen lymphocytes (TAA-T) with Nivolumab response, change from baseline at year one. Response will be assessed by imaging using the Lugano criteria. Response is defined as any patient who does not progress on this study, including patients with active disease who achieve Complete Metabolic Response (CMR)/Complete Response (CR), Partial Metabolic Response (PMR)/ Partial Response (PR), or No Metabolic Response(NMR)/Stable Disease (SD) by PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Boyu Hu, MD, Principal Investigator — UTAH
Locations (1):
- Utah University School of Medicine/Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Dave H, Terpilowski M, Mai M, Toner K, Grant M, Stanojevic M, Lazarski C, Shibli A, Bien SA, Maglo P, Hoq F, Schore R, Glenn M, Hu B, Hanley PJ, Ambinder R, Bollard CM. Tumor-associated antigen-specific T cells with nivolumab are safe and persist in vivo in relapsed/refractory Hodgkin lymphoma. Blood Adv. 2022 Jan 25;6(2):473-485. doi: 10.1182/bloodadvances.2021005343. PMID 34495306